CLINICAL TRIAL: NCT03117959
Title: A Randomized Control Trial Comparing an Anatomical Axis Aligned and Conventional Mechanical Axis Total Knee Arthroplasty Using Patient-Specific Instrumentation
Brief Title: TKA Using Patient-Specific Instrumentation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no longer RCT - same surgical technique and implant used
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Gavin Wood, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SURG-290-14; 6011807 (Other: Queen's University TRAQ system)
Record Dates: First submitted 2014-04-07; First posted 2017-04-18 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stryker Triathlon Custom Fit Knee (Placebo Comparator): implanted in standard fashion
  Interventions: Device: Stryker Triathlon Custom Fit Knee
- Stryker shape match (Experimental): no longer RCT
  Interventions: Device: Stryker ShapeMatch Technology

INTERVENTIONS:
Device: Stryker ShapeMatch Technology — Will use this patient-specific guide for alignment with Stryker Triathlon Custom Fit Knee.
  Arms: Stryker shape match
Device: Stryker Triathlon Custom Fit Knee
  Arms: Stryker Triathlon Custom Fit Knee

SUMMARY:
The purpose of our study is to determine if anatomic/kinematic total knee arthroplasties (TKAs) are superior to mechanical axis-referenced TKAs with respect to determinants of gait functionality, patient satisfaction and other objective tests of knee function as a potential indicator of long-term prosthesis outcomes. To our knowledge there has not been any literature comparing TKAs using the kinematic and mechanical axes with respect to gait analysis. A single study has compared gender-specific TKAs and found that there is no difference with respect to determinants of gait when using these prostheses (Thomsen et al, 2012), but again this study was not based on referencing off of the anatomical/kinematic axis of the knee. Our group is hoping that the small variability that may be detectable with the precision of gait analysis may be used as a predictor of future prosthesis outcome measures.

DETAILED DESCRIPTION:
The reference standard for total knee replacement or total knee arthroplasty (TKA) has historically been based on a 2-dimensional "mechanical axis" of the knee which surgically creates a joint line parallel to the ground. This is based on the idea that this alignment will evenly distribute the stress on the prosthesis, thus improving the wear characteristics and longevity of the replacement. More recent studies have shown that TKAs with greater than 3 degree deviation (in either valgus or varus) from this previously accepted ideal does not convey a survival benefit over a 15 year period. This is not to say that alignment does not play a role in survivorship as gross deviation from neutral does result in earlier implant failure, but a simple 2-D model may not be the ideal approach to TKAs. With the developments and improvements in patient-specific technology (or patient-specific instrumentation (PSI)), our ability to create TKAs that reproduce the patient's original anatomic or kinematic alignment in 3-Dimensions has dramatically improved. Early research with respect to function and survivorship has shown that PSIs are at least equivalent when compared to conventional TKAs. Some studies have also suggested improvements with respect to shorter operating times, less blood loss and increased range of motion. Most of the current PSI TKA literature has placed an emphasis on the technology's effect on TKA alignment or to show that it is bioequivalent with respect to range of motion or early prosthesis survivorship when compared to conventional TKAs. Although a single study using PSIs (Howell et al., 2013) has shown improvement in Oxford Knee Scores when comparing patients preoperatively to postoperatively, to our knowledge there is no research done to directly compare the functional knee scores between a mechanically-aligned and anatomically aligned TKA. This randomized control trial will compare these two approaches using implants from the same manufacturer and also hope to identify more subtle functional differences using power testing and gait analysis, in addition to assessing other perioperative outcomes such as blood loss, hospital stay duration and operative time.

ELIGIBILITY:
Inclusion Criteria:

* Aged = 50-75
* BMI = 20 - 40
* Preoperative ability to perform certain gait tasks/skills
* No previous knee surgery or injury on either limb
* No neuromuscular disease or neurologic disease
* ASA of 1-2

Exclusion Criteria:

* below age 50 and/or above age 75
* BMI less than 20 or greater than 40
* ASA of 3 or higher

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
gait analysis | 12 months
  Treadmill walk

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Wood, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No